CLINICAL TRIAL: NCT04934839
Title: Instrumental Analysis of Walking in People With Osseointegrated Prostheses for Lower Extremity Amputation: Comparative Evaluation With Traditional Socket Prostheses
Acronym: AStrO-OI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: ASST Gaetano Pini-CTO (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24X101
Record Dates: First submitted 2021-05-31; First posted 2021-06-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Lower Extremity Amputation
Keywords: Lower extremity amputation; Osseointegrated prostheses; Learned non-use; Rehabilitation; Walking; Gait analysis; Split-belt treadmill; Balance; Osseointegration

STUDY DESIGN:
Intervention Model Description: Osseointegration for lower limb amputation is a rare procedure. Therefore, a convenience sample of patients will be enrolled. Efforts will be made to match the participants with controls, fitted with conventional socket prosthesis, by age, gender, height and weight without the prosthesis, prosthetic side, and type of prosthesis, but an exact matching is not considered a strict requirement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with osseointegrated prostheses (Experimental): Patients with an osseointegrated prosthesis following a lower limb amputation
  Interventions: Diagnostic Test: Test of standing balance (Equitest System). Test of walking in tied and split conditions on a force-sensorized split-belt treadmill.
- Patients with socket prostheses (Experimental): Patients with a socket-mounted prosthesis following a lower limb amputation
  Interventions: Diagnostic Test: Test of standing balance (Equitest System). Test of walking in tied and split conditions on a force-sensorized split-belt treadmill.

INTERVENTIONS:
Diagnostic Test: Test of standing balance (Equitest System). Test of walking in tied and split conditions on a force-sensorized split-belt treadmill. — Tests of standing balance will be performed using the EquiTest System posturographic platform. Individuals will be requested to perform three tasks within the EquiTest battery: Sensory Organization test, Motor Control test backward/forward, Adaptation Test upward/downward.
  Gait analysis will be performed on a force sensorized split-belt treadmill. Participants will walk at increasing velocities from 0.2 m/s to the highest sustainable velocity in tied-belt condition. Velocity will be increased by 0.1 m/s every 20 consecutive strides.
  During gait analysis in the split-belt condition, participants will walk for 30 seconds with both belts at 0.4 m/s. Then, the velocity of the belt under the prosthetic limb will be increased to 1.2 m/s. After 6 minutes, the velocity of the faster belt will be restored at 0.4 m/s for 6 more minutes. Different combinations of velocities could be tested based on the patients' characteristics, maintaining a ratio of 3:1 between the velocities of the 2 belts.

SUMMARY:
The currently accepted standard for rehabilitation and mobility following amputation is a socket-mounted prosthesis. Osseointegration is an alternative method that has gradually gained greater acceptance in the last 30 years. It is defined as a procedure in which a metal implant is directly anchored to the residual bone, attached to a prosthetic limb using a transcutaneous connector.

The advantages of osseointegrated prostheses over conventional socket prostheses include stable fixation, significant increases in walking ability, range of motion and control of the prosthesis, and health-related quality of life. Moreover, bodyweight distribution results more similar to physiological conditions.

No formal consensus exists for osseointegration surgery. However, based on the positive clinical experience, surgeons currently indicate this surgery for those patients who show poor tolerance of socket prostheses.

The present study investigates neuro-physiologic and mechanical parameters of walking and balance in patients with lower limb amputation and osseointegrated prostheses and in matched patients with traditional socket prostheses to highlight strengths and weaknesses of the alternative technique with respect to the present standard of care.

The primary endpoint is the investigation of the neurologic and mechanic adaptation in terms of a) kinematic and dynamic segmental analysis of walking and transfer of the body center of mass during walking; b) capacity to retain balance in response to different conditions of oscillation, tilt, and translation of a posturographic platform.

The secondary endpoint is investigating of adaptation to walking on a split-belt treadmill mounted on force sensors with the belts running at different velocities.

We hypothesize that:

* the deficit in joint power of the prosthetic limb is associated with a phenomenon of "learned non-use" both in balance and during gait. This behavior looks automatic and unconscious. It consists of the under recruitment of the impaired side as a form of unconscious protection, which is adopted when the contralateral side may be exploited to carry out the function;
* the joint power provided by the prosthetic limb may increase both by increasing treadmill velocity and by walking in split-belt modality with the prosthetic limb on the faster belt;
* an "after-effect" will be evidenced after the split-belt walking test when the two belts will return to the same velocity; patients with osseointegrated prostheses and patients with socket prostheses may show different behaviors in the adaptation to split-belt walking and the following post-adaptation, as a result of the residual proprioception of the amputated limb.

Results from the present study will allow:

* the identification of the possible advantages in walking and balance symmetry in patients with osseointegrated prostheses with respect to patients with socket prostheses;
* the estimate of the sample size for future experimental protocols and new rehabilitative programs.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower extremity amputation;
* age > 18 years;
* amputation-adjusted Body Mass Index between 18 and 25;
* ability to understand the instructions;
* ability to wittingly sign the informed consent form.

Exclusion Criteria:

* other previous knee injuries or major surgical interventions at the lower limbs;
* comorbidities, such as neurological conditions, vascular diseases, or diseases of orthopedic, cardiac, or pulmonary origin;
* cancer disease in the site under examination;
* other neurological pathologies with impact on balance and gait.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Joint power | Day 1
  Joint kinematics will be recorded during walking through an optoelectronic method as per the Davis anthropometric model. The 3D displacement of the markers will be captured using 8 near-infrared stroboscopic cameras. Joint power will be computed through the spatiotemporal synchronization of ground reaction force vectors and the joint centers of rotation. The sagittal plane, only, will be considered for the analysis. Hip, knee, and ankle joint power will be computed as the product of joint torque and joint rotation speed. Power will be defined as positive or generated when the joint moment and rotation speed share the same directions (i. e., when agonist muscles are contracting while shortening), as negative or absorbed otherwise. Positive work will be computed as the integral of the generated (positive) power over time.

SECONDARY OUTCOMES:
Kinetic energy of the center of mass during walking | Day 1
  Changes in kinetic energy during walking due to the forward (Ekf), lateral (Ekl), and vertical (Ekv) velocity will be computed.
Energy of the center of mass during walking due to vertical motion | Day 1
  Changes in gravitational potential energy (Ep), and changes of the mechanical energy due to the vertical motion, Ev = Ekv+Ep, will be computed.
Total mechanical energy of the center of mass during walking | Day 1
  Changes in total mechanical energy (Etot = Ekf+Ekl +Ev) will be computed.
Recovery of mechanical energy, R | Day 1
  The amount of recovery of mechanical energy, R, due to the passive exchange between Ekf, Ev and Ekl, during walking, will be computed according to the equation R = (Wf + Wv + Wl - Wext)/(Wf + Wv + Wl) × 100, where Wf for Ekf, Wv for Ev, Wl for Ekl and Wtot for Etot represents the corresponding work values calculated as the sum of the positive increments of these energy values during one step.
SOT score | Day 1
  The patient's task is to maintain an upright stance during three 20 s trials under six different conditions, including movements of the platform and the visual surround 'tuned' with the individual's sagittal oscillation. The SOT score will be calculated by comparing the sagittal oscillation of the body's center of mass (COM) to the maximal sagittal oscillation. The score is averaged across the six conditions (range 0-100. The higher the score, the lower the oscillation).
MCT score | Day 1
  The patient's capacity to recover upright stance when the platform suddenly shifts forward or backward, thus causing the subject to lean back or forward with respect to the ground. The score is the latency between the onset of translation and the rise of a compensatory torque. Average latency between legs, repetitions and stimulus amplitude (36 values overall) is computed. The score is given in ms (the lower, the better).
ADT score | Day 1
  The patient's capacity to minimize body sway when the platform suddenly tilts upward or downward, thus causing the body to lean backward or forward with respect to the ground, respectively. A non-dimensional parameter from a 'sway-energy function' is calculated. The function provides an 'energy' parameter derived from the root mean square of speed and acceleration of the position of the centre of pressure on the force plate during the tilt (range 0 to infinite, the lower, the better).

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tesio, MD, Professor, Principal Investigator — Istituto Auxologico Italiano
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, Milan, MI
  - ASST Gaetano Pini-CTO, Milan

IPD SHARING:
Plan to Share IPD: Yes